CLINICAL TRIAL: NCT04191551
Title: The GAstric Precancerous Conditions Study
Acronym: GAPS
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-45077; NCI-2020-13776 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Intestinal Metaplasia of Gastric Mucosa; Helicobacter Pylori Infection; Atrophic Gastritis
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Blood Gastric specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Precursor lesions: Subjects with precursor lesions detected on endoscopy.

SUMMARY:
Gastric cancer afflicts 27,000 Americans annually and carries a dismal prognosis. One reason for poor outcomes is late diagnosis, as the majority of gastric cancers in the United States are diagnosed at a relatively advanced stage where curative resection is unlikely. Gastric precursors (such as atrophic gastritis and intestinal metaplasia) are precancerous changes to the stomach mucosa which increases risk for subsequent gastric cancer.

The Gastric Precancerous Conditions Study (GAPS) is an observational study of patients at elevated risk for gastric cancer. Investigators seek to recruit patients from endoscopy unit of Stanford Health Care, a large academic network of hospitals and clinics serving Northern California. Investigators will recruit patients who are both symptomatic (e.g. dyspepsia) and asymptomatic (e.g. referred for screening), and individuals both with known precursor lesions (such as intestinal metaplasia) or at high risk for carrying precursor lesions. A component of the study is long-term follow-up of individuals with gastric precursors. This is to understand their risk factors for histologic progression and regression. During both index and subsequent endoscopies, the study team will collect biospecimens (e.g. blood, saliva, gastric tissue).

ELIGIBILITY:
Inclusion Criteria: Subjects between the ages of 35 and 84, who are undergoing outpatient endoscopy for the following indications are eligible: abdominal pain, dyspepsia, iron deficiency anemia, Helicobacter assessment, surveillance of suspected or known intestinal metaplasia, evaluation for family history of gastric cancer

Exclusion Criteria:

* Cannot give consent
* Have history of gastric surgery
* Have history of solid tumor or bone marrow transplant
* Platelet Count < 70 or international normalized ratio > 1.5

Ages: 35 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Histologic Progression or Regression Assessed by OLGA Score | at least 24 months after enrollment
  Histologic progression or regression will be evaluated using the Operative Link on Gastritis Assessment (OLGA) score. This score stages the severity of atrophic gastritis based on histological findings.
Histologic Progression or Regression Assessed by OLGIM Score | at least 24 months after enrollment
  Histologic progression or regression will be assessed using the Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) score. This score stages the extent of intestinal metaplasia.
Development of Dysplasia | at least 24 months after enrollment
  The presence or absence of dysplasia will be assessed as an indicator of histologic progression.
Development of Carcinoma | at least 24 months after enrollment
  The presence or absence of carcinoma will be assessed to evaluate disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Huang, MD, Principal Investigator — Stanford University; Joo Ha Hwang, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided